CLINICAL TRIAL: NCT03656341
Title: Foot Self-care in Older Adults Without Diabetes
Brief Title: Foot Self-care in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jennifer O'Connor, PhD student, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011705
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Foot
Keywords: foot care; older adults; senior center; self-management; self-care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2 Feet 4 Life (Experimental): Intervention group will receive one hour intervention weekly for four consecutive weeks. Outcomes will be measured at baseline (before the intervention), immediately after the intervention (1 month), three months post-intervention, and six months post-intervention
  Interventions: Behavioral: 2 Feet 4 Life
- True control group (No Intervention): Will complete the same four assessment visits as the intervention group.
- Bias control group (No Intervention): Will complete outcome assessments at baseline and the final assessment.

INTERVENTIONS:
Behavioral: 2 Feet 4 Life — 2 Feet 4 Life consists of four weekly group intervention sessions of one hour each. 2 Feet 4 Life includes self-management teaching, interactive lecture, and group activities, including instruction and demonstration of routine foot care. The program includes education regarding appropriate footwear and how to find it, evidenced based practices on hygiene, skin care and self-care of the lower extremities, nail trimming and filing, and care of common foot problems.
  Arms: 2 Feet 4 Life

SUMMARY:
This pilot study will make a preliminary evaluation of the efficacy of 2 Feet 4 Life, a foot care self-management program, on foot care knowledge, foot care self-efficacy, foot care behaviors, and foot pain in community dwelling older adults without diabetes mellitus.

DETAILED DESCRIPTION:
One in three older adults have foot problems such as bunions, corns, calluses, foot pain, or nail disorders, but those problems are often ignored or overlooked until they threaten mobility or quality of life. With proper self-management, skin and nail problems can be addressed before they become severe; however, older adults without diabetes are not routinely informed of self-management techniques unless they consult a specialist. Targeting a foot care self-management program to community-dwelling older adults without diabetes may not only enhance foot function and preserve independence but also reach older adults with limited healthcare access.

Study participants will be 24 nondiabetic older adults recruited from two Midwestern community senior centers. One community center will be randomized to receive the intervention, 2 Feet 4 Life, the other will be a true control group receiving no intervention. The 2 Feet 4 Life foot care self-management program is based on Social Cognitive Theory and will be delivered in four weekly, one-hour group sessions. The program includes self-management teaching, interactive lecture, and group activities, including instruction, demonstration, and practice of routine foot care. In addition to usual lecture and handouts, 2 Feet 4 Life will rely on group interaction, practice opportunities, and the provision of foot care supplies so participants can perform foot care at home. Program topics include appropriate foot hygiene and footwear, identification and treatment of common foot problems, demonstration of proper foot care with opportunities for practice and instructor feedback, and guidance in obtaining appropriate footwear.

Outcome measures will be assessed pre-intervention, immediately post-intervention, three months post-intervention, and six months post-intervention. This will be the first study to test a nurse run, community-based, foot care self-management program for non-diabetic older adults.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* legally competent to sign informed consent
* willing to participate in the study

Exclusion Criteria:

* self-reports of diabetes
* non-traumatic amputation
* legal blindness.
* demonstrated inability to see and remove dot stickers on the feet
* active ingrown toenails
* absent pedal pulses
* poor sensation as defined by the inability to feel more than 3 of 10 foot sites touched with a microfilament
* regular visits to a healthcare professional for foot care
* score of <2 on the mental status screener.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Foot Self-Care Knowledge Questionnaire | Baseline, one month, three months, six months
  0-11 scale with higher numbers indicating more knowledge
Foot Care Confidence Scale | Baseline, one month, three months, six months
  12-60 scale with greater scores indicating greater self-efficacy
Nottingham Assessment of Functional Foot Care | Baseline, one month, three months, six months
  Scale of 0-87 with higher scores revealing more appropriate foot self-care
Manchester Foot Pain and Disability INdex | Baseline, one month, three months, six months
  0-34 scale with higher scores indicating more pain and disability

SECONDARY OUTCOMES:
Foot Health Score | Baseline, one month, three months, six months
  Scale 0-90 provider assessment of foot problems. Higher score indicate more severe foot problems and greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer O'Connor, Principal Investigator — University of Missouri-Columbia
Locations (2):
- United States (2):
  - Broken Arrow Seniors, Broken Arrow, Oklahoma
  - Owasso Community Center, Owasso, Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baba M, Duff J, Foley L, Davis WA, Davis TM. A comparison of two methods of foot health education: the Fremantle Diabetes Study Phase II. Prim Care Diabetes. 2015 Apr;9(2):155-62. doi: 10.1016/j.pcd.2014.05.004. Epub 2014 Jun 12. PMID 24929632
- [Background] Barr EL, Browning C, Lord SR, Menz HB, Kendig H. Foot and leg problems are important determinants of functional status in community dwelling older people. Disabil Rehabil. 2005 Aug 19;27(16):917-23. doi: 10.1080/09638280500030506. PMID 16096244
- [Background] Castillo A, Giachello A, Bates R, Concha J, Ramirez V, Sanchez C, Pinsker E, Arrom J. Community-based Diabetes Education for Latinos: The Diabetes Empowerment Education Program. Diabetes Educ. 2010 Jul-Aug;36(4):586-94. doi: 10.1177/0145721710371524. Epub 2010 Jun 10. PMID 20538970
- [Background] Garrow AP, Papageorgiou AC, Silman AJ, Thomas E, Jayson MI, Macfarlane GJ. Development and validation of a questionnaire to assess disabling foot pain. Pain. 2000 Mar;85(1-2):107-13. doi: 10.1016/s0304-3959(99)00263-8. PMID 10692609
- [Background] Haas L, Maryniuk M, Beck J, Cox CE, Duker P, Edwards L, Fisher EB, Hanson L, Kent D, Kolb L, McLaughlin S, Orzeck E, Piette JD, Rhinehart AS, Rothman R, Sklaroff S, Tomky D, Youssef G; 2012 Standards Revision Task Force. National standards for diabetes self-management education and support. Diabetes Care. 2014 Jan;37 Suppl 1(Suppl 1):S144-53. doi: 10.2337/dc14-S144. No abstract available. PMID 24357210
- [Background] Mickle KJ, Munro BJ, Lord SR, Menz HB, Steele JR. Cross-sectional analysis of foot function, functional ability, and health-related quality of life in older people with disabling foot pain. Arthritis Care Res (Hoboken). 2011 Nov;63(11):1592-8. doi: 10.1002/acr.20578. PMID 22034121
- [Background] Senussi, M., Lincoln, N., & Jeffcoate, W. (2011). Psychometric properties of the Nottingham Assessment of Functional Footcare (NAFF). International Journal of Therapy and Rehabilitation, 18(6), 330-334. https://doi.org/10.12968/ijtr.2011.18.6.330
- [Background] Snider KT, Seffinger MA, Ferrill HP, Gish EE. Trainer-to-student ratios for teaching psychomotor skills in health care fields, as applied to osteopathic manipulative medicine. J Am Osteopath Assoc. 2012 Apr;112(4):182-7. PMID 22522517
- [Background] Stolt M, Suhonen R, Puukka P, Viitanen M, Voutilainen P, Leino-Kilpi H. Foot health and self-care activities of older people in home care. J Clin Nurs. 2012 Nov;21(21-22):3082-95. doi: 10.1111/j.1365-2702.2012.04223.x. Epub 2012 Jul 27. PMID 22835017
- [Background] Waxman R, Woodburn H, Powell M, Woodburn J, Blackburn S, Helliwell P. FOOTSTEP: a randomized controlled trial investigating the clinical and cost effectiveness of a patient self-management program for basic foot care in the elderly. J Clin Epidemiol. 2003 Nov;56(11):1092-9. doi: 10.1016/s0895-4356(03)00197-5. PMID 14615000

DOCUMENTS (1):
  • Informed Consent Form (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/41/NCT03656341/ICF_000.pdf